CLINICAL TRIAL: NCT01816685
Title: The Effect of Peri-operative Continuous Positive Airway Pressure (CPAP) on Postoperative Delirium in a Population at High-risk for Obstructive Sleep Apnea (OSA)
Brief Title: Effect of CPAP on Postoperative Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00041457
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Sleep Apnea, Obstructive; Delirium
MeSH Terms: conditions — Sleep Apnea, Obstructive; Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- CPAP (Experimental): Patients in the CPAP group will be instructed to wear an autotitrating positive airway pressure (APAP) device any time they sleep prior to surgery and on postoperative days 0, 1, and 2.
  Interventions: Device: CPAP
- Routine Care (No Intervention)

INTERVENTIONS:
Device: CPAP
  Arms: CPAP

SUMMARY:
Patients with a medical condition known as obstructive sleep apnea may be at increased risk of delirium following surgery. This study loans autotitrating CPAP machines to randomly-selected patients who are at high-risk for obstructive sleep apnea with the goal of preventing post-operative delirium.

DETAILED DESCRIPTION:
Patients undergoing elective knee and hip replacements will be prospectively enrolled. These surgical procedures all have an expected length of stay > 3 days. Immediately following enrollment, patients will be randomized to receive CPAP or routine peri-operative care. Patients in the CPAP group will be instructed to wear an autotitrating positive airway pressure (APAP) device any time they sleep prior to surgery and on postoperative days 0, 1, and 2.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and above
* Scheduled for an elective knee or hip replacement
* Ability to speak English and give informed consent
* At risk for obstructive sleep apnea as defined by a STOP-BANG score > 2

Exclusion Criteria:

* History of psychiatric or neurologic illness that would confound delirium assessment
* Severe tracheal or lung disease
* Contraindications to face-mask CPAP
* Treated OSA

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krystal, MD, Principal Investigator — Department of Psychiatry, Duke University Medical Center
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Derived] Evans JL, Nadler JW, Preud'homme XA, Fang E, Daughtry RL, Chapman JB, Attarian D, Wellman S, Krystal AD. Pilot prospective study of post-surgery sleep and EEG predictors of post-operative delirium. Clin Neurophysiol. 2017 Aug;128(8):1421-1425. doi: 10.1016/j.clinph.2017.05.004. Epub 2017 May 17. PMID 28618293

RESULTS

PARTICIPANT FLOW:
Groups:
- CPAP: Patients in the continuous positive airway pressure (CPAP) group will be instructed to wear an autotitrating positive airway pressure (APAP) device any time they sleep prior to surgery and on postoperative days 0, 1, and 2.
- Routine Care: Routine care will be provided to the participant.
Period: Overall Study
Arm/Group | CPAP | Routine Care
Started | 68 | 67
Completed | 58 | 56
Not Completed | 10 | 11
Not completed — Lost to Follow-up | 7 | 9
Not completed — Surgery Cancelled | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP | Routine Care | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 65 [60 to 70] | 65 [59 to 71] | 65 [60 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 32 | 68
  Male | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Presence of Postoperative Delirium
Description: Assessments for delirium were made on postoperative day 2 using the Delirium Rating Scale-Revised-98 (DRS-R-98) diagnostic and assessment tool. The DRS-R-98 is a 16-item clinician-rated scale that consists of a severity score (maximum score 39, minimum 0) made up of items that can be used for repeated serial measurements and a total scale score (maximum score 46, minimum 0) that includes the severity score plus three diagnostic items (7 additional possible points) used for initial ratings. Items represent symptoms that are rated on a scale of 0 to 3 points, with text descriptions for each point. Higher scores on the scale represents a larger number of delirium symptoms or increased severity of those symptoms.
Time Frame: Postoperative day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CPAP | Routine Care
Number analyzed (Participants) | 58 | 56
units on a scale
  DRS-R-98 severity score | 4.8 (4.3) | 5.1 (4.3)
  DRS-R-98 total score | 7.8 (6.4) | 8.1 (6)

2. Primary Outcome: Presence of Postoperative Delirium
Description: Assessments for delirium were made on postoperative day 2 using the Confusion Assessment Method (CAM) Diagnostic Algorithm. This binary tool identifies the presence or absence of delirium
Time Frame: Postoperative day 2
Measure: Number; unit: participants
Arm/Group | CPAP | Routine Care
Number analyzed (Participants) | 58 | 56
participants | 12 | 9

ADVERSE EVENTS:
Groups:
- CPAP: Patients in the CPAP group will be instructed to wear an autotitrating positive airway pressure (APAP) device any time they sleep prior to surgery and on postoperative days 0, 1, and 2.
  CPAP
Arm/Group | CPAP | Routine Care
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/56
Other Adverse Events (participants affected / at risk) | 0/58 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes